CLINICAL TRIAL: NCT03393494
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Perrigo's Adapalene/BP Gel to Galderma's Epiduo (Adapalene/BP) Gel, and Both Treatments to a Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: Bioequivalence Study of Two Treatments in the Treatment of Acne Vulgaris on the Face
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-17-008
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Perrigo active (Experimental): Test product
  Interventions: Drug: Adapalene and Benzoyl Peroxide Topical Gel
- Reference active (Active Comparator): RLD product
  Interventions: Drug: Epiduo Topical Product
- Perrigo placebo (Placebo Comparator): placebo product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene and Benzoyl Peroxide Topical Gel — Test product
  Arms: Perrigo active
Drug: Epiduo Topical Product — RLD product
  Arms: Reference active
Drug: Placebo — Placebo gel
  Arms: Perrigo placebo

SUMMARY:
To compare the safety and efficacy of Perrigo's product to an FDA approved product for the treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

1. Signed IRB approved written informed consent/assent
2. 12 to 40 years of age, inclusive.
3. Clinical diagnosis of facial acne vulgaris with an inflammatory lesion (papules and pustules) count of 20-50, inclusive and a non-inflammatory (open and closed comedones) lesion count of 25-100 inclusive and no more than 2 nodulocystic lesions (e.g., nodules and cysts) including those present on the nose.
4. Baseline Investigator's Global Assessment Score of 3 (moderate) or 4 (severe) on a severity scale of 0 to 4.
5. Females of child bearing potential (excluding women who are surgically sterilized (tubal ligation or bilateral oophorectomy or hysterectomy) or post-menopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day1(Baseline), must be willing to use an acceptable form of birth control during the study.

Exclusion Criteria:

1. Pregnant, breastfeeding or planning a pregnancy within the period of their study participation period.
2. Presence of more than 2 facial Nodulocystic lesions.
3. Presence of any other facial skin condition that, in the Investigator's opinion, might interfere with acne vulgaris diagnosis and/or evaluations
4. Any uncontrolled, chronic or serious disease or medical condition that would prevent participation in a clinical trial, or, in judgment of the investigator, would put the subject at undue risk or might confound the study assessments
5. Excessive facial hair that would interfere with the diagnosis or assessment of acne vulgaris.
6. History of unresponsiveness to topical adapalene and/or benzoyl peroxide therapy.
7. Currently using any product containing adapalene and/or benzoyl peroxide and/or belonging to the same family.
8. History of hypersensitivity or allergy to adapalene, benzoyl peroxide, retinoids and/or any ingredient in the study medication.
9. Use of medications known to exacerbate acne
10. Start or change within 3 months (90 days) of Visit 1 and throughout the study
11. Use of medicated make-up throughout the study and significant change in the use of consumer products within 30 days (1 month) of study entry and throughout the study
12. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements.
13. Subjects who in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 825 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consultants, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Adapalene and Benzoyl Peroxide Topical Gel
- Reference Product: Epiduo Topical Gel
- Placebo Product: Placebo gel
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 329 | 331 | 165
Completed | 261 | 256 | 140
Not Completed | 68 | 75 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perrigo Active | Reference Active | Perrigo Placebo | Total
Number analyzed (Participants) | 329 | 331 | 165 | 825
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 160 | 161 | 76 | 397
  Between 18 and 65 years | 169 | 170 | 89 | 428
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 129 | 69 | 315
  Male | 212 | 202 | 96 | 510
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 126 | 120 | 53 | 299
  Not Hispanic or Latino | 203 | 211 | 112 | 526
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 4
  Asian | 13 | 6 | 4 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 51 | 48 | 30 | 129
  White | 241 | 256 | 122 | 619
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 21 | 19 | 9 | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in the Papules and Pustules Lesion Count
Time Frame: Day 1 to week 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of lesion change
Arm/Group | Perrigo Active | Reference Active | Perrigo Placebo
Number analyzed (Participants) | 202 | 218 | 120
percentage of lesion change | 68.18 (28.96) | 63.56 (31.57) | 50.72 (35.12)
Statistical Analysis 1: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — provides 85% power of success; Fieller's method; Equivalence ratio = 107, 90% CI 2-sided [97.8 to 112.2]

2. Primary Outcome: Mean Percent Change From Baseline in the Open and Closed Comedones Lesion Count
Description: Per protocol population
Time Frame: Day 1 to week 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of lesion change
Arm/Group | Perrigo Active | Reference Active | Perrigo Placebo
Number analyzed (Participants) | 202 | 218 | 120
percentage of lesion change | 62.75 (28.09) | 60.78 (33.73) | 43.45 (36.30)
Statistical Analysis 1: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — provides 85% power of success; p = 0.05, Fieller's method; Equivalence ratio = 104, 90% CI 2-sided [94.1 to 108.5]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Perrigo Active | Reference Active | Perrigo Placebo
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/331 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/331 | 2/165
Other Adverse Events (participants affected / at risk) | 0/329 | 0/331 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perrigo Active (N=329) | Reference Active (N=331) | Perrigo Placebo (N=165)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03393494/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03393494/SAP_000.pdf